CLINICAL TRIAL: NCT06249061
Title: A Randomised Controlled Feasibility Trial of Oral Sodium Bicarbonate for the Prevention of Labour Dystocia
Brief Title: Oral Sodium Bicarbonate for the Prevention of Labour Dystocia
Acronym: Labour-Aide
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liz Darling (Other)
Collaborators: Trillium Health Partners (Other); London Health Sciences Centre (Other); Oak Valley Health (Other)
Responsible Party: Sponsor-Investigator, Liz Darling, Associate Professor, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REB 4424
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Labour Dystocia
Keywords: dystocia; labor; sodium bicarbonate
MeSH Terms: conditions — Dystocia | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Sodium Bicarbonate (Experimental): Those in the intervention group will be encouraged to sip a solution of sodium bicarbonate (1 imperial teaspoon (~5g) of sodium bicarbonate dissolved into 250ml of water; if the entire 250mL is consumed, another 1 imperial teaspoon (~5g) of sodium bicarbonate dissolved in 250mL of water will be provided to the patient) throughout labour with other drinks as desired. All other care will remain the same.
  Interventions: Dietary Supplement: oral sodium bicarbonate
- Usual Care (No Intervention): Those in the usual care group will be encouraged to sip fluids of their choice throughout labour as they would normally be encouraged to do. All other care will remain the same.

INTERVENTIONS:
Dietary Supplement: oral sodium bicarbonate — Those in the oral sodium bicarbonate intervention group will be encouraged to sip a solution of 1 imperial teaspoon (~5g) of sodium bicarbonate dissolved into 250ml of water throughout labour with other drinks. If the first solution is fully consumed, a second solution will be prepared and offered. Thus, each participant can receive a maximum dose of 2 imperial teaspoons (~10g) of sodium bicarbonate.
  Other Names: Bicarbonate De Soude Usp by Laboratoire Atlas Inc
  Arms: Oral Sodium Bicarbonate

SUMMARY:
Sodium bicarbonate is often used by athletes to improve their muscle's ability to contract and power their activity. It works by decreasing the risk of lactic acid build-up, which causes cramping and fatigue. Some research suggests that using sodium bicarbonate in labour could help to improve the ability of the uterus to contract, helping to prevent labour dystocia (stalled or slow progress in labour). This could ultimately increase the chance of spontaneous vaginal delivery. This research is being done to investigate whether drinking sodium bicarbonate (commonly known as baking soda) dissolved in water as a hydration drink could benefit women in labour and increase the chance of a vaginal birth. In order to answer this question, pregnant people from London, Markham and Mississauga midwifery practices are being recruited to participate in this study. Participants will be randomly assigned to one of two groups when they are admitted to hospital in labour. One group will be asked to drink normal fluids of their choice while they are in labour (usual care). The second group will be asked to consume a drink made of baking soda and water, as well as normal fluids of their choice. Mode of birth and the use of birth interventions will be compared between the two groups. Infant outcomes will be compared to ensure that the use this drink in labour is safe. A risk of consuming sodium bicarbonate is gastrointestinal disturbance. The number of people who reported gastrointestinal upset will also be compared between the two groups. If this study shows that those who drank sodium bicarbonate in labour had an increased chance of vaginal birth and that it is safe, this low-cost, low-risk treatment has the potential to reduce birth interventions for pregnant people and their babies.

DETAILED DESCRIPTION:
Sodium bicarbonate is used by athletes to improve muscle contractility and decrease the risk of lactic acid build-up. A moderately sized efficacy study suggests that these proposed effects may be beneficial for nulliparous women in labor to maintain efficiency of labour contractions. Sodium bicarbonate may be useful for improving the contractility of the uterus, helping to prevent labour slowing (dystocia) and ultimately increasing the rate of spontaneous vaginal deliveries. Large scale randomized controlled trials (RCTs) are necessary to determine the effectiveness of sodium bicarbonate for prevention of labour dystocia.

This is an unblinded, open-label, two-arm (treatment vs. usual care control), feasibility RCT evaluating oral sodium bicarbonate for the prevention of labour dystocia for nulliparous midwifery clients at two centres. This study will be conducted with the primary aim of determining feasibility for a full-scale RCT to answer the question: are nulliparous women in midwifery care who receive oral sodium bicarbonate as a hydration drink in labour more or less likely to fail to achieve spontaneous vaginal birth compared to women who drink fluids of their choice? This feasibility study will take place at 4 hospitals in Ontario (Mississauga Hospital, Credit Valley Hospital, Markham Stouffville Hospital, London Health Sciences Centre) and will aim to recruit as many participants as possible during an 8-month period.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant,
2. Nulliparous,
3. Cephalic presenting,
4. Live, singleton fetus,
5. Planning hospital birth,
6. Under the care of a midwife
7. In spontaneous active labour (with or without cervical ripening), and
8. Greater than or equal to (≥) 37weeks, and 0 days gestation. There is no maximum gestation, so long as the labour was spontaneous

Exclusion Criteria:

1. Planning caesarean birth,
2. Hypertension requiring treatment,
3. Diabetes or gestational diabetes requiring pharmacological treatment,
4. On a low sodium diet,
5. Use of illicit drugs in pregnancy, or
6. Unable to provide informed consent or understand instructions on ingestion of the substance
7. Oxytocin induction of labour, or
8. Oxytocin augmentation of labour prior to randomisation

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a full-scale RCT | 8 months of recruitment
  Feasibility will be determined by assessing recruitment, compliance, participant retention, side effects, completeness of data, participant satisfaction and facilitators and barriers to study implementation.

SECONDARY OUTCOMES:
Failure to achieve a spontaneous vaginal birth | At the time of birth
  Composite of Caesarean section and assisted vaginal birth

CONTACTS AND LOCATIONS:
Overall Officials: Liz Darling, PhD, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: No